CLINICAL TRIAL: NCT02579187
Title: Efficacy of Local Delivery of MicroRNAs and MicroRNA Inhibitors in Promoting Osteogenesis and Modulating Local Inflammation: A Pilot Clinical Trial Using the Tooth Socket Model
Brief Title: MicroRNA and MicroRNA Inhibitors Socket Study, Pilot Clinical Trial
Status: Withdrawn | Phase: Phase 1 | Type: Interventional
Why Stopped: withdrawn study from IRB
Sponsor: Gustavo Avila-Ortiz DDS, MS, PhD (Other)
Responsible Party: Sponsor-Investigator, Gustavo Avila-Ortiz DDS, MS, PhD, DDS, University of Iowa
Organization: University of Iowa (Other)
Allocation: Randomized | Model: Parallel | Masking: Single | Purpose: Health Services Research
Other Study IDs: 201607780
Record Dates: First submitted 2015-10-12; First posted 2015-10-19 (Estimated); Last update posted 2019-07-17 (Actual); Status verified 2019-07

CONDITIONS: Tooth Extraction Status Nos
MeSH Terms: interventions — Tooth Extraction; Anesthesia; Blood Specimen Collection; Phlebotomy; Videotape Recording

STUDY DESIGN:
Who Masked: Participant
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: Yes | FDA-regulated Device: No | US Export: No

ARMS (4):
- control group (Placebo Comparator): CBCT scan limited to the dental arch that includes the study site will be obtained. All subjects will receive local infiltrative anesthesia, following which minimally invasive tooth extraction will be performed. After tooth extraction clinical measurements of the site will also be obtained and recorded for both groups (i.e. keratinized mucosa width, horizontal ridge width, facial and lingual bone thickness). A biodegradable sponge (type I bovine collagen) to stabilize the blood clot will be placed.The site will be stabilized with a simple external, cross mattress suture. Blood , wound fluid, and saliva samples will be taken periodicallly. In addition, photos/videos, periapical xrays and PVS impressions will be obtained.
  Interventions: Procedure: tooth extraction; Radiation: CBCT scan; Drug: Anesthesia; Other: clinical measurements; Drug: Biodegradable sponge (type I bovine collagen); Procedure: cross mattress suture; Procedure: Blood; Other: Photos/videos; Procedure: Wound fluid; Procedure: saliva; Radiation: periapical xray; Other: PVS impression
- Experimental group 1 (Active Comparator): CBCT scan limited to the dental arch that includes the study site will be obtained. All subjects will receive local infiltrative anesthesia, following which minimally invasive tooth extraction will be performed. After tooth extraction clinical measurements of the site will also be obtained and recorded for both groups (i.e. keratinized mucosa width, horizontal ridge width, facial and lingual bone thickness). 10µg of pSil-miR200c plasmids in a biodegradable sponge (type I bovine collagen) will be locally delivered. The site will be stabilized with a simple external, cross mattress suture. Blood, wound fluid, and saliva samples will be taken periodicallly. In addition, photos/videos, periapical xrays and PVS impressions will be obtained.
  Interventions: Procedure: tooth extraction; Radiation: CBCT scan; Drug: Anesthesia; Other: clinical measurements; Drug: 10µg of pSil-miR200c; Procedure: cross mattress suture; Procedure: Blood; Other: Photos/videos; Procedure: Wound fluid; Procedure: saliva; Radiation: periapical xray; Other: PVS impression
- Experimental group 2 (Active Comparator): CBCT scan limited to the dental arch that includes the study site will be obtained. All subjects will receive local infiltrative anesthesia, following which minimally invasive tooth extraction will be performed. After tooth extraction clinical measurements of the site will also be obtained and recorded for both groups (i.e. keratinized mucosa width, horizontal ridge width, facial and lingual bone thickness). 10µg of PMIS miR200a plasmids in a biodegradable sponge (type I bovine collagen) will be locally delivered. The site will be stabilized with a simple external, cross mattress suture. Blood, wound fluid, and saliva samples will be taken periodicallly. In addition, photos/videos, periapical xrays and PVS impressions will be obtained.
  Interventions: Procedure: tooth extraction; Radiation: CBCT scan; Drug: Anesthesia; Other: clinical measurements; Procedure: cross mattress suture; Drug: 10µg of PMIS miR200a plasmids; Procedure: Blood; Other: Photos/videos; Procedure: Wound fluid; Procedure: saliva; Radiation: periapical xray; Other: PVS impression
- Experimental group 3 (Active Comparator): CBCT scan limited to the dental arch that includes the study site will be obtained. All subjects will receive local infiltrative anesthesia, following which minimally invasive tooth extraction will be performed. After tooth extraction clinical measurements of the site will also be obtained and recorded for both groups (i.e. keratinized mucosa width, horizontal ridge width, facial and lingual bone thickness). 5µg of pSil-miR200c and 5µg of PMIS miR200a plasmids in a biodegradable sponge (type I bovine collagen) will be locally delivered. The site will be stabilized with a simple external, cross mattress suture. Blood, wound fluid, and saliva samples will be taken periodicallly. In addition, photos/videos, periapical xrays and PVS impressions will be obtained.
  Interventions: Procedure: tooth extraction; Radiation: CBCT scan; Drug: Anesthesia; Other: clinical measurements; Procedure: cross mattress suture; Drug: 5µg of pSil-miR200c and 5µg of PMIS miR200a; Procedure: Blood; Other: Photos/videos; Procedure: Wound fluid; Procedure: saliva; Radiation: periapical xray; Other: PVS impression

INTERVENTIONS:
Procedure: tooth extraction — The study tooth will be removed
Radiation: CBCT scan — a CBCT scan limited to the dental arch that includes the study side will be obtained
Drug: Anesthesia — all subjects will receive local infiltrative anesthesia, prior to extraction of the tooth
  Other Names: local infiltrative anesthesia
Other: clinical measurements — After tooth extraction, clinical measurements of the site will be obtained and recorded (keratinized mucosa width, horizontal ridge width, facial and lingual bone thickness
Drug: Biodegradable sponge (type I bovine collagen) — control group subjects will receive a biodegradable sponge (type I bovine collagen) to stabilize the clot
  Other Names: Bovine collagen
  Arms: control group
Drug: 10µg of pSil-miR200c — subjects in the experimental group will receive a 10µg of pSil-miR200c plasmids in a biodegradable sponge (type I bovine collagen) to stabilize the clot
  Other Names: pSil-miR-200C plasmids
  Arms: Experimental group 1
Procedure: cross mattress suture — The site will be stabilized with a simplet external, cross mattress suture
Drug: 10µg of PMIS miR200a plasmids — subjects in the experimental group will receive a 10µg of PMIS miR200a plasmids in a biodegradable sponge (type I bovine collagen) to stabilize the clot
  Other Names: PMIS miR200a plasmids
  Arms: Experimental group 2
Drug: 5µg of pSil-miR200c and 5µg of PMIS miR200a — subjects in the experimental group will receive a 5µg of pSil-miR200c and 5µg of PMIS miR200a plasmids in a biodegradable sponge (type I bovine collagen) to stabilize the clot
  Other Names: 5µg of pSil-miR200c and 5µg of PMIS miR200a plasmids
  Arms: Experimental group 3
Procedure: Blood — Subjects will have venipuncture performed to obtain a small blood sample (approx. 2 ml) to assess for miR-200c and PMIS-miR-200a expression and liver function (AST, ALT, bilirubin levels)
  Other Names: venipuncture
Other: Photos/videos — subjects will have photos and/or videos of the extraction site and/or implant taken at each visit.
Procedure: Wound fluid — a small sample of wound fluid will be obtained from the extraction site in a minimally invasive manner using a paper point at 1, 2, 3 & 4 weeks post extraction
Procedure: saliva — approximately 2 mls of saliva will be obtained in a minimally invasive manner at the time of extraction and at 14 weeks post extraction.
Radiation: periapical xray — periapical xrays will be obtained at screening, 16 weeks and at 12 month followup time point
Other: PVS impression — PVS impressions will be taken to plan the implant placement surgery. This will be done at the screening visit and also at 14 weeks post extraction.

SUMMARY:
To evaluate the efficacy of locally delivering plasmid DNAs encoding microRNAs, and/or microRNA inhibitors, in the promotion of osteogenesis and modulation of the inflammatory response on the basis of different clinical, radiographic, histologic and biomolecular outcomes in post-extraction socket defects in humans.

DETAILED DESCRIPTION:
The purpose of this study is to evaluate the efficacy of locally delivering plasmid DNAs encoding microRNAS and/or microRNA inhibitors, a naturally occurring microRNA molecule, in the promotion of bone formation and attenuation of local inflammation in a tooth socket model in humans.

Patients requiring tooth extractions and future tooth replacement therapy with a dental implant will be eligible for the study. Recruited subjects will be randomly assigned to either a control (tooth extraction and 10µg empty vector in bovine collagen sponge) or one of 3 experimental groups:

* Experimental group 1: Tooth extraction and bovine collagen sponge containing 10µg of pSil-miR200c
* Experimental Group 2: Tooth extraction and bovine Collagen sponge containing 10µg of PMIS miR200a
* Experimental Group 3: Tooth extraction and bovine Collagen sponge containing 5µg of pSil-miR200c and 5µg of PMIS miR200a

Subjects will be clinically re-evaluated at 1, 2, 3 and 4 weeks. In each one of these visits, a fluid sample will be obtained from the healing site in a minimally invasive manner to assess local biomolecular profiles. Blood samples will be drawn at 1, 2, 3, 4 and 14 week visits to assess for miR-200c and PMIS-miR 200a expression and liver function. Photos and/or videos will also be obtained. A CBCT scan and a saliva sample (approx. 2 ml) will also be obtained at baseline and at 14 weeks to assess bone volume and intraoral biomolecular profiles, respectively.

Implant placement surgery will be performed at 16 weeks from the time of tooth extraction. A bone core biopsy will be harvested at this time for histologic analysis. A periapical radiograph (small dental x-ray image) will be obtained at baseline (before tooth extraction) and at 14 weeks (prior to implant placement) to assess bone height changes.

Follow-up visits will occur at 6 months and 12 months post implant at which time measurements and photos will be taken.

ELIGIBILITY:
INCLUSION CRITERIA

* Age: 25 to 65 years.
* Gender: No restriction.
* Subjects must require a single-rooted tooth extraction (Tooth deemed as periodontally, endodontically and/or restoratively hopeless).
* Subjects must be able and willing to follow instructions related to the study procedures.
* Subjects must have read, understood and signed an informed consent form.

EXCLUSION CRITERIA

* Reported allergy or hypersensitivity to any of the products to be used in the study.
* Severe hematologic disorders, such as leukemia.
* Active severe infectious diseases that may compromise normal healing.
* Liver or kidney dysfunction/failure.
* Currently under cancer treatment or history of cancer of any kind.
* Subjects who have a long-term history of oral bisphosphonate use (i.e. 4 years or more).
* Subjects with a history of IV bisphosphonates.
* Subjects with uncontrolled diabetes.
* Subjects with severe metabolic bone diseases, such as Paget's disease of bone, will be excluded.
* Pregnant women or nursing mothers.
* Smokers: Within 6 months of study onset.
* Concomitant medications: Subjects on concomitant drug therapy for systemic conditions, such as antibiotics or patient taking non-steroidal anti-inflammatory (NSAID) agents that may affect the outcomes of the study will not be included in the study. Subjects taking biologics or disease modifying agents will also be excluded. Occasional, short-term use (7-14 days) of analgesics or common cold medications is permitted.
* Any other non-specified reason that from the point of views of the investigators will make a candidate not a suitable subject for the study (e.g. limited mouth opening).

Ages: 25 Years to 65 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Enrollment: 0 (Actual)
Dates: Start 2025-12-31 (Estimated); Primary Completion 2030-09 (Estimated); Study Completion 2030-09 (Estimated)

PRIMARY OUTCOMES:
Percent of mineralized tissue upon histomorphometric analysis of bone core biopsies | at 16 weeks postoperatively
  compared using exact Wilcoxon rank sum tests

SECONDARY OUTCOMES:
Bucco-lingual width changes of the alveolar ridge (in mm) | up to 16 weeks postoperatively
  Fisher's exact tests will be used to compare the treatment groups
Mid-buccal height changes of the alveolar ridge (in mm) | up to 16 weeks postoperatively
  compared using exact Wilcoxon rank sum tests
Mid-lingual height changes of the alveolar ridge (in mm) | up to 16 weeks postoperatively
  compared using exact Wilcoxon rank sum tests
Volumetric reduction of the alveolar ridge (in cc) via CBCT scan analyses | at 16 weeks postoperatively
  compared using exact Wilcoxon rank sum tests
Expression of different biomarkers (VEGF, PDGF, TGF-b, IL-1b, TNF-a) in wound fluid expressed in pg/ml | up to 4 weeks postoperatively
  compared using exact Wilcoxon rank sum tests

CONTACTS AND LOCATIONS:
Overall Officials: Brad Amendt, MS, Study Director — UIowa College of Dentistry
Locations (1):
- UIowa, Iowa City, Iowa, United States

IPD SHARING:
Plan to Share IPD: Undecided